CLINICAL TRIAL: NCT03134781
Title: The Effects of a Novel Hybrid Exercise Training Program on Body Composition, Body Weight and Energy Balance in Sedentary Overweight/Obese Women
Brief Title: Hybrid Exercise Training for Weight Loss
Acronym: DoIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DoIT-UTH
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Circuit-based High Intensity Interval Training; Body Composition; Resting Metabolic Rate; Habitual Physical Activity; Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): Participated only in measurements at baseline, at 20 weeks and at 40 weeks.
  Interventions: Behavioral: Control - No training
- Training (Experimental): Participated in a supervised 40-week DoIT workout exercise training program and in measurements at baseline, at 20 weeks and at 40 weeks.
  Interventions: Behavioral: DoIT workout
- Training-Detraining (Experimental): Participated in a supervised 20-week DoIT workout exercise training program and then entered a 20-week detraining period. They also participated in measurements at baseline, at 20 weeks and at 40 weeks.
  Interventions: Behavioral: DoIT workout - Detraining

INTERVENTIONS:
Behavioral: DoIT workout — A hybrid small-group (5-10 women/session) training modality, that combines interval training, resistance exercise and functional training and performed according to a periodized model of exercise prescription as an alternative approach for weight management. FFIT was performed 3 times/week with 48 hours recovery between sessions for 40 weeks.
  Arms: Training
Behavioral: DoIT workout - Detraining — A hybrid small-group (5-10 women/session) training modality, that combines interval training, resistance exercise and functional training, performed according to a periodized model of exercise prescription for a 20-week period (3 times/week). Immediately after a 20-week detraining period (no training was performed) was followed.
  Arms: Training-Detraining
Behavioral: Control - No training — No training was performed during a 40-week period. Participation only in measurements.
  Arms: Control

SUMMARY:
In this study the investigators utilized a novel hybrid HIIT (high intensity interval training) exercise training approach, the Hybrid Interval Training (DoIT) workout that combines interval training, resistance exercise training and functional training in order to test the hypothesis that DoIT will be able to: i) reduce body mass, ii) improve body composition and iii) alter energy balance, of previously inactive, overweight/obese women.

DETAILED DESCRIPTION:
In a controlled randomized, two-group, repeated measures design, 65 healthy, sedentary, premenopausal overweight or obese women were randomly assigned to one of three groups: (a) a control group (C, N=21) that participated only in measurements, (b) a training group (TR, N=14) that participated in a supervised 40-week DoIT workout exercise training program and (c) a training-detraining group (TRD, N=14). During the first 20 weeks, TR and TRD followed exactly the same training protocol. At the end of this period, TR continued training for 20 more weeks whereas TRD terminated training for 20 weeks (detraining). Anthropometric, metabolic, daily nutritional intake, habitual physical activity and performance measurements were performed in all groups at baseline, at 20 weeks and 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* (a) were sedentary (<7,500 steps/day; VO2max <30 ml/kg/min), b) premenopausal women aged 30-45 years, c) were overweight or obese class 1 (BMI=25-34.9 kg/m2), d) were non-smokers for ≥6 months before the study, e) not following a diet intervention or using nutritional supplements/medications before (≥6 months) and during the study, f) had no weight loss greater >10% of body mass ≤6 months before the study, g) participated in ≥80% of total exercise sessions, and h) had no symptoms of depression.

Exclusion Criteria:

* a) a recent febrile illness, b) history of muscle lesion, c) lower limb trauma, d) signs, symptoms or diagnosis of serious health complications or physical disability or other medical condition compromising safe participation in exercise training.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in body mass | At baseline, at 20 weeks and at 40 weeks.
Change in body mass index | At baseline, at 20 weeks and at 40 weeks.
Change in waist circumference | At baseline, at 20 weeks and at 40 weeks.
Change in hip circumference | At baseline, at 20 weeks and at 40 weeks.
Change in waist-to-hip ratio | At baseline, at 20 weeks and at 40 weeks.
Change in body fat. | At baseline, at 20 weeks and at 40 weeks.
  Body fat assessed by whole-body dual-energy X-ray absorptiometry (DXA).
Change in fat mass | At baseline, at 20 weeks and at 40 weeks.
  Fat mass assessed by whole-body dual-energy X-ray absorptiometry (DXA).
Change in fat-free mass | At baseline, at 20 weeks and at 40 weeks.
  Fat-free mass assessed by whole-body dual-energy X-ray absorptiometry (DXA).
Change in resting metabolic rate | At baseline, at 20 weeks and at 40 weeks.
  Measured using a portable open-circuit indirect calorimeter with a ventilated hood system.
Change in exercise-induced caloric expenditure. | At baseline, at 20 weeks and at 40 weeks.
  Measured using a portable indirect calorimetry system

SECONDARY OUTCOMES:
Change in maximal strength (1RM) | At baseline, at 20 weeks and at 40 weeks.
  Measured bilaterally on a horizontal leg press.
Change in maximal oxygen consumption (VO2max) | At baseline, at 20 weeks and at 40 weeks.
  Assessed by a portable open-circuit spirometry system.
Change in blood lactate concentration | Pre-exercise, during the exercise and post-exercise at baseline, at 20 weeks and at 40 weeks.
Change in habitual physical activity | At baseline, at 20 weeks and at 40 weeks.
  Seven-day habitual physical activity was assessed by accelerometry
Change in dietary intake | At baseline, at 20 weeks and at 40 weeks.
  Assessed using 7-day diet recalls

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Biochemistry Laboratory, School of Physical Education & Sports Sciences, University of Thessaly, Trikala, Karies, Greece

REFERENCES:
- [Result] Batrakoulis A, Jamurtas AZ, Georgakouli K, Draganidis D, Deli CK, Papanikolaou K, Avloniti A, Chatzinikolaou A, Leontsini D, Tsimeas P, Comoutos N, Bouglas V, Michalopoulou M, Fatouros IG. High intensity, circuit-type integrated neuromuscular training alters energy balance and reduces body mass and fat in obese women: A 10-month training-detraining randomized controlled trial. PLoS One. 2018 Aug 23;13(8):e0202390. doi: 10.1371/journal.pone.0202390. eCollection 2018. PMID 30138475
- [Result] Batrakoulis A, Loules G, Georgakouli K, Tsimeas P, Draganidis D, Chatzinikolaou A, Papanikolaou K, Deli CK, Syrou N, Comoutos N, Theodorakis Y, Jamurtas AZ, Fatouros IG. High-intensity interval neuromuscular training promotes exercise behavioral regulation, adherence and weight loss in inactive obese women. Eur J Sport Sci. 2020 Jul;20(6):783-792. doi: 10.1080/17461391.2019.1663270. Epub 2019 Sep 16. PMID 31478436
- [Result] Batrakoulis A, Tsimeas P, Deli CK, Vlachopoulos D, Ubago-Guisado E, Poulios A, Chatzinikolaou A, Draganidis D, Papanikolaou K, Georgakouli K, Batsilas D, Gracia-Marco L, Jamurtas AZ, Fatouros I. Hybrid neuromuscular training promotes musculoskeletal adaptations in inactive overweight and obese women: A training-detraining randomized controlled trial. J Sports Sci. 2021 Mar;39(5):503-512. doi: 10.1080/02640414.2020.1830543. Epub 2020 Oct 15. PMID 33054601
- [Result] Batrakoulis A, Jamurtas AZ, Draganidis D, Georgakouli K, Tsimeas P, Poulios A, Syrou N, Deli CK, Papanikolaou K, Tournis S, Fatouros IG. Hybrid Neuromuscular Training Improves Cardiometabolic Health and Alters Redox Status in Inactive Overweight and Obese Women: A Randomized Controlled Trial. Antioxidants (Basel). 2021 Oct 12;10(10):1601. doi: 10.3390/antiox10101601. PMID 34679738
- [Derived] 2020 NSCA Research Abstracts. J Strength Cond Res. 2021 Apr 1;35(4):e3-e288. doi: 10.1519/JSC.0000000000003877. No abstract available. PMID 33752224